CLINICAL TRIAL: NCT02959814
Title: Diagnostic Accuracy of On-line Quantitative Flow Ratio. Functional Assessment by Virtual Online Reconstruction (The FAVOR II Europe-Japan Study)
Brief Title: Diagnostic Accuracy of On-line Quantitative Flow Ratio (QFR). FAVOR II Europe-Japan
Acronym: FAVOR II EJ
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Niels Ramsing Holm, Research associate, M.D., Aarhus University Hospital Skejby
Other Study IDs: 1-10-72-219-16
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve; Quantitative Coronary Analysis; Stable coronary artery disease; Angina pectoris
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: QFR (observational) — QFR assessment by Medis Suite, Medis medical imaging B.V., The Netherlands

SUMMARY:
Quantitative Flow Ratio (QFR) is a novel method for evaluating the functional significance of coronary stenosis. QFR is assessed by calculation of the pressure in the vessel based on two angiographic projections. The purpose of the FAVOR II study is to evaluate the diagnostic accuracy of on-line QFR compared to 2D Quantitative Coronary Angiography (QCA) with FFR as gold standard.

DETAILED DESCRIPTION:
Background:

Patients at high risk of having one or more coronary stenosis are evaluated routinely by invasive coronary angiography (CAG). Lesions are often quantified by QCA, but fractional flow reserve is increasingly used to assess functional significance of identified stenosis. FFR is assessed during CAG by advancing a wire with a pressure transducer towards the stenosis and measure the ratio in pressure between the two sides of the stenosis during medical induced maximum blood flow (hyperaemia).

The solid evidence for FFR evaluation of coronary stenosis and the relative simplicity in performing the measurements have supported adoption of an FFR based strategy in many centers but the need for interrogating the stenosis by a pressure wire, the cost of the wire, and the drug inducing hyperaemia limits more widespread adoption.

Quantitative Flow Ratio is a novel method for evaluating the functional significance of coronary stenosis by calculation of the pressure drop in the vessel based on two angiographic projections.

The FAVOR I study (Tu et al.), showed promising results for core laboratory QFR analysis in selected patients.

The purpose of the FAVOR II study is to evaluate the feasibility and diagnostic precision of in-procedure QFR during CAG in comparison to QCA with FFR as gold standard for physiological lesion evaluation.

Hypothesis: QFR has superior sensitivity and specificity for detection of functional significant lesions in comparison to QCA with FFR as gold standard

Methods: Prospective, observational, multicenter study with inclusion of 310 patients.

Patients with indication for FFR are enrolled. At least two angiographic projections are acquired during resting conditions. QFR is calculated in-procedure using the Medis Suite application and simultaneously to the operator performing the FFR measurement. The QFR observer is blinded to the FFR measurement.

QFR is reassessed off-line by the Interventional Coronary Imaging Core Laboratory, Aarhus University, Denmark, blinded to FFR and in-procedure QFR results.

FFR is assessed by core laboratory reading, blinded to QFR results. All data are entered and stored in a protected and logged trial management system (TrialPartner, Aarhus University, Denmark).

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris or secondary evaluation of stenosis after acute MI
* Age > 18 years
* Able to provide signed informed consent
* Angiographic inclusion criteria:
* Indication for FFR in at least one stenosis:
* Diameter stenosis of 30%-90% by visual estimate
* Reference vessel size > 2 mm in stenotic segment by visual estimate

Exclusion Criteria:

* Myocardial infarction within 72 hours
* Severe asthma or severe chronic obstructive pulmonary disease
* Severe heart failure (NYHA≥III)
* S-creatinine>150µmol/L or GFR<45 ml/kg/1.73m2
* Allergy to contrast media or adenosine
* Atrial fibrillation
* Angiographic exclusion criteria:

Lesion specific

* Below 30% and above 90% diameter stenosis by visual estimate.
* Reference size of vessel below 2 mm by visual estimation.
* Ostial LMCA lesions
* Ostial RCA lesions
* Distal LMCA lesions in combination with proximal Cx lesions
* Other bifurcation stenosis with lesions on both sides of a major shift (>1mm) in reference diameter Angiographic quality
* Poor image quality precluding contour detection
* Good contrast filling not possible
* Severe overlap of stenosed segments
* Severe tortuosity of target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable angina pectoris admitted for coronary angiography due to high risk of significant coronary stenosis
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niels R. Holm, M.D., Principal Investigator — Aarhus University Hospital, Denmark
Locations (10):
- Aarhus University Hspital, Aarhus N, Denmark
- Institut Cardiovasculaire Paris Sud Massy, Massy, France
- Germany (2):
  - Elizabeth Krankenhaus Essen, Essen
  - Universitätsklinikum Gießen, Giessen
- Italy (3):
  - Azienda ospedaliera Sant'Anna e S. sebastiano di Caserta, Caserta
  - Azienda Ospedaliero-Universitaria di Ferrara, University of Ferrara, Ferrara
  - Ospedale dell'Angelo di Mestre, Mestre
- Gifu Heart Center, Gifu, Japan
- HagaZiekenhuis, The Hague, Netherlands
- Golden Jubilee National Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Derived] Westra J, Andersen BK, Campo G, Matsuo H, Koltowski L, Eftekhari A, Liu T, Di Serafino L, Di Girolamo D, Escaned J, Nef H, Naber C, Barbierato M, Tu S, Neghabat O, Madsen M, Tebaldi M, Tanigaki T, Kochman J, Somi S, Esposito G, Mercone G, Mejia-Renteria H, Ronco F, Botker HE, Wijns W, Christiansen EH, Holm NR. Diagnostic Performance of In-Procedure Angiography-Derived Quantitative Flow Reserve Compared to Pressure-Derived Fractional Flow Reserve: The FAVOR II Europe-Japan Study. J Am Heart Assoc. 2018 Jul 6;7(14):e009603. doi: 10.1161/JAHA.118.009603. PMID 29980523

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Paired QFR, FFR and 2D-QCA: Patients with stable angina pectoris or secondary evaluation of stenosis after acute MI reffered to invasive coronary angiography (ICA). ICA revealed at least one lesion with 30-90 % diameter stenosis with indication for fractional flow reserve (FFR). No lesions were excluded by the FFR, 2D-QCA nor angiographic criteria
Period: Overall Study
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Started | 329 (22-02-2017)
Completed | 272 (17-10-2017)
Not Completed | 57
Not completed — Excluded based on diagnostic angiography | 16
Not completed — Excluded based on anatomical criteria | 2
Not completed — Protocol Violation | 7
Not completed — FFR not measured | 2
Not completed — In-procedure QFR not computed | 6
Not completed — Excluded by FFR core-lab | 24

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 196
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity: Proportion of Patients With Positive QFR of FFR Positive Patients (True Positives) Compared to Proportion of Patients With Positive Percentual Diameter Stenosis (DS%) Assessed by 2D QCA of FFR Positive Patients (True Positives)
Description: Positive FFR is defined as FFR≤0.80. Positive QFR is defined as QFR≤0.80. Positive DS% is defined as DS% > 50%
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Proportion
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Proportion
  2D-QCA | 0.442 [0.345 to 0.543]
  QFR | 0.865 [0.784 to 0.924]

2. Primary Outcome: Specificity: Proportion of Patients With Negative QFR of FFR Negative Patients (True Negatives) Compared to Proportion of Patients With Negative DS% Assessed by 2D QCA of FFR Negative Patients (True Negatives)
Description: Negative FFR is defined as FFR>0.80. Negative QFR is defined as QFR>0.80. Negative DS% is defined as DS% ≤ 50%.
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Proportion
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Proportion
  2D-QCA | 0.765 [0.703 to 0.820]
  QFR | 0.869 [0.816 to 0.911]

3. Secondary Outcome: Percentage of Patients With Successful QFR in Patients With Successful FFR (Feasibility)
Time Frame: 1 hour
Population: Patients with successful FFR Measurement before Exclusion based on missing QFR and/or 2D-QCA
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Measured FFR: Patients with succesfull FFR measurement
Arm/Group | Patients With Measured FFR
Number analyzed (Participants) | 302
Participants | 296

4. Secondary Outcome: Proportion of Patients With Positive QFR of FFR Positive Patients (True Positives) (Sensitivity)
Description: Positive FFR is defined as FFR≤0.80. Positive QFR is defined as QFR≤0.80
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Proportion
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Proportion | 0.865 [0.784 to 0.924]

5. Secondary Outcome: Proportion of Patients With Negative QFR of FFR Negative Patients (True Negatives) (Specificity)
Description: Negative FFR is defined as FFR>0.80. Negative QFR is defined as QFR>0.80
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Proportion
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Proportion | 0.869 [0.816 to 0.911]

6. Secondary Outcome: Proportion of Patients With Positive FFR (True Positives) of Patients With Positive QFR (Positive Predictive Value)
Description: Positive FFR is defined as FFR≤0.80. Positive QFR is defined as QFR≤0.80
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Proportion
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Proportion | 0.763 [0.676 to 0.836]

7. Secondary Outcome: Proportion of Patients With Negative FFR (True Negatives) of Patients With Negative QFR (Negative Predictive Value)
Description: Negative FFR is defined as FFR>0.80. Negative QFR is defined as QFR>0.80
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Proportion
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Proportion | 0.930 [0.885 to 0.961]

8. Secondary Outcome: Diagnostic Performance of QFR in Comparison to FFR Reported as Positive and Negative Likelihood Ratio
Description: Positive likelihood ratio is defined as sensitivity/(1-specificity). Negative likelihood ratio is defined as (1-sensitivty)/specificity
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Ratio
  Negative likelihood ratio | 0.16 [0.09 to 0.25]
  Positive likelihood ratio | 6.60 [4.62 to 9.37]

9. Secondary Outcome: Diagnostic Grey Zone Calculation. QFR Limits for Achieving 95% Sensitivity and Specificity in Comparison to FFR
Description: QFR limits to yield 95% sensitivity and specificity. The QFR limits are identified by Area under the receiver operating curve analysis.
  QFR limits are defined as the numerical QFR ratios (0-1.00).
Time Frame: 1 hour
Measure: Number; unit: Ratio
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Ratio
  95% limit for sensitivity | 0.77
  95% limit for specificity | 0.87

10. Secondary Outcome: Diagnostic Accuracy of TIMI-flow Based QFR in Comparison to 2D QCA (>50% Diameter Stenosis)
Description: Comparison of proportion of participants correctly classified by QFR and 2D QCA using FFR as reference standard.
  Diagnostic accuracy is defined as (true positives + false negatives) / (true positives+false positives+true negatives+false negatives).
  Positive FFR is defined as FFR≤0.80. Positive QFR is defined as QFR≤0.80. Negative FFR is defines as FFR>0.80. Negative QFR is defines as QFR>0.80. Positive 2D QCA is defined as 2D-QCA % percent diameter stenosis >50. Negative 2D QCA is defined as 2D-QCA % diameter stenosis≤50.
Time Frame: 1 hour
Measure: Number; unit: Proportion
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Proportion
  TIMI-FLOW based QFR | 0.868
  2D-QCA | 0.659

11. Secondary Outcome: Participants With Myocardial Infarction (Number of Patients)
Description: Peri-procedural myocardial infarction
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Participants | 0

12. Secondary Outcome: All-cause Mortality (Number of Patients)
Description: Peri-procedural mortality
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Participants | 0

13. Secondary Outcome: Time to FFR
Description: Time from starting preparations to do FFR (e.g. ordering assistants to prepare pressure wire, adenosine infusion etc.) to FFR value is obtained and drift has been verified to be within the prespecified limits
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Minutes | 7.0 [5.0 to 10.0]

14. Secondary Outcome: Time to QFR After Receiving Angiographic Images
Description: Time from first image evaluation on QFR computer until TIMI frame count based QFR value is obtained
Time Frame: 1 hour
Measure: Mean (Inter-Quartile Range); unit: Minutes
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Minutes | 5.0 [3.5 to 6.1]

15. Secondary Outcome: Contrast Use
Description: Volume of contrast for total procedure
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
mL | 120 (76)

16. Secondary Outcome: Fluoroscopy Time
Description: Fluoroscopy time for total procedure
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
Number analyzed (Participants) | 272
Minutes | 9.8 (7.2)

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Patients With Paired QFR, FFR and 2D-QCA
All-Cause Mortality (participants affected / at risk) | 0/329
Serious Adverse Events (participants affected / at risk) | 0/329
Other Adverse Events (participants affected / at risk) | 0/329

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT02959814/Prot_SAP_000.pdf